CLINICAL TRIAL: NCT04766853
Title: Verification of the Efficacy / Safety of the Intratympanic Drug Delivery Vehicle for Treating Intractable Hearing Loss (pilot Study)
Brief Title: Verification of the Efficacy/safety of the Intratympanic Drug Delivery for Hearing Loss
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-1812-128-997
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-07

CONDITIONS: Hearing Loss, Sudden; Hearing Loss, Ototoxic; Hearing Loss, Noise-Induced; Meniere Disease
Keywords: Hearing loss; Drug Delivery; Dexamethasone; Hyaluronic Acid; Intratympanic injection
MeSH Terms: conditions — Hearing Loss, Sudden; Hearing Loss; Hearing Loss, Noise-Induced; Meniere Disease | interventions — Dexamethasone; Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexamethasone+Saline (Active Comparator)
  Interventions: Drug: Dexamethasone
- Dexamethasone+Hyaluronic Acid (Experimental)
  Interventions: Drug: Dexamethasone; Drug: Hyaluronic acid

INTERVENTIONS:
Drug: Dexamethasone — Dexamethasone 5mg/ml
Drug: Hyaluronic acid — Hyaluronic Acid 20mg/2ml
  Arms: Dexamethasone+Hyaluronic Acid

SUMMARY:
This study is a prospective, randomized pilot study. To verify an efficacy and safety of the Intratympanic drug delivery vehicle, patients who have not responded to the existing standard treatment will be enrolled. Hearing test, endoscopy of tympanic membrane and CT scans will be conducted after intratympanic treatment for evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Sudden hearing loss, ototoxic hearing loss, noise-induced hearing loss, meniere's disease patients with 25dB HL in pure tone audiometry
* Patients whose hearing has not been restored after standard treatment
* Patients do not participate in clinical trials within 6 months

Exclusion Criteria:

* Patients with retrocochlear lesion
* Patients with history of hypersensitivity to the ingredients of this drug
* Patients with end-stage renal disease, end-stage liver disease, cardiovascular surgery, progressive brain tumor, progressive palsy and progressive stroke, etc. severe brain disease or cancer.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-07-22 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2024-07-19 (Actual)

PRIMARY OUTCOMES:
Verification of tympanic membrane with endoscopy (Safety) | 3-4 weeks after intratympanic injection
  Confirming healing time of perforation and inflammation
Confirmation of inflammation and drug with CT imaging (Durability) | 1 day and/or 1 weeks after intratympanic injection
  Checking a time duration of drug in middle and inner ear
Valuation of hearing threshold with Pure tone audiometry (Efficacy) | 3-4 weeks after intratympanic injection
  Verifying therapeutic effect of intratympanic drug delivery vehicle

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea